CLINICAL TRIAL: NCT04636398
Title: Development and Pilot Test of an mHealth Interactive Education and Social Support Intervention for Improving Postnatal Health - Phase 1
Brief Title: Postnatal mHealth Intervention Development
Acronym: MESSAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Los Angeles (Other); Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Indraprastha Institute of Information Technology Delhi (Other); Survival for Women and Children Foundation (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R21HD101786 (NIH); R21HD101786 (NIH)
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Results first posted 2022-08-19 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Health Attitude; Knowledge, Attitudes, Practice; Postpartum Depression; Acceptability of Health Care
MeSH Terms: conditions — Behavior; Depression, Postpartum; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Non-randomized quasi-experimental exploratory study. All small groups will receive the same intervention which is exposure to a variety of intervention modalities (3 main modalities: information delivery, facilitation strategy, text management).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MESSAGE mHealth group intervention (Experimental): Participants in the one arm will be exposed to the mHealth group intervention. As this is a pilot developmental study, the participants will be exposed to various strategies for information delivery (live presentation at a scheduled time versus voice recording accessible at any time), discussion facilitation (heavily managed with request to speak vs. natural discussion participation), and text communication management (moderator-facilitated vs. group-led).
  Interventions: Behavioral: MESSAGE - mHealth intervention

INTERVENTIONS:
Behavioral: MESSAGE - mHealth intervention — A group-based moderated six-week intervention with didactic, discussion, and text communication components.

SUMMARY:
This study is a six-week exploratory developmental phase (phase 1) of a larger project to develop an mHealth intervention targeting health education and social support for Indian women in the postnatal period. Phase 1 of the trial exposes study participants to various intervention modalities and seeks to understand their experiences and perspectives on these using mixed-methods. Results from this trial will inform modifications to the intervention to be tested in Phase 2.

DETAILED DESCRIPTION:
Most mHealth interventions for maternal and child health (MCH) in low and middle-income countries, including India, have focused on unidirectional and non-interactive approaches, primarily text messaging. However, ample evidence suggests that provider-led, interactive educational programming and social support are key for improving health behaviors and outcomes. Thus innovative mHealth approaches that promote interactive education and facilitate social support have great potential to improve MCH outcomes. The two-phase development of MeSSSSage will include Phase 1: exploratory development on functions and platforms and Phase 2: a mixed-methods randomized pilot study using a factorial design of specific intervention functions and platforms confirmed in Phase 1. Study activities described herein are associated with Phase 1. The study's specific aim is: To develop optimal intervention functions, processes, and mHealth platforms for education and peer support among postnatal women in rural India. In Phase 1, the investigators will explore potential interactive education and peer support group intervention functions (education, emotional support, instrumental support, referrals, linkages, follow-up on postnatal visits), processes (group interactions; frequency, length and timing of groups; engagement opportunities, participant profiles) and mHealth delivery platforms (voice, text chat, app options, interaction features). This six-week developmental component will include up to four groups (n=48; 12 per group) to assess different modalities and functions. The investigators will ascertain women's preferences for functions, processes, and platform features using survey and in-depth interviews (IDIs), and capture levels of engagement via back-end data. This process will also inform the intervention's health information content. Findings will be used to formalize the group mobile intervention details to be examined in Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Postnatal (within 2 weeks)
* 18+ years old

Exclusion Criteria:

* Women below 18 years of age
* Women with high risk pregnancies
* Women who delivered preterm, suffer severe maternal complications or they or their baby are otherwise sick in the first week

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison El Ayadi, ScD, Principal Investigator — University of California, San Francisco; Nadia G Diamond-Smith, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Post Graduate Institute for Medical Education and Research (PGIMER), Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MESSAGE mHealth Group Intervention
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MESSAGE mHealth Group Intervention
Number analyzed (Participants) | 29
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 25 [24 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  India | 29
Personal smartphone [Number; unit: participants] | 17
Educational attainment [Count of Participants; unit: Participants]
  Illiterate | 3
  Primary | 2
  Higher primary | 4
  Secondary | 3
  Senior secondary | 11
  Graduation | 3
  Post-Graduation | 3

OUTCOME MEASURES:

1. Primary Outcome: Satisfied or Very Satisfied About Their Overall Intervention Experience
Description: Proportion of participants reporting to be "satisfied" or "very satisfied" with their overall intervention experience, assessed through a five-point Likert scale at six weeks.
Time Frame: 6 weeks
Population: We were unable to recruit an additional person to reach our target sample size of 30 within the time frame and criteria required for the group-oriented intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | MESSAGE mHealth Group Intervention
Number analyzed (Participants) | 29
Participants | 29

ADVERSE EVENTS:
Time Frame: 6 weeks of intervention participation
Arm/Group | MESSAGE mHealth Group Intervention
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT04636398/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT04636398/SAP_001.pdf
  • Informed Consent Form (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT04636398/ICF_002.pdf